CLINICAL TRIAL: NCT04766476
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 1b Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BMS-963272 in Participants With Nonalcoholic Fatty Liver Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, and Drug Levels of BMS-963272 in Participants With Nonalcoholic Fatty Liver Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB006-025
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: BMS-963272; Liver Fibrosis; Nonalcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis (NASH); Phase 1b
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Treatment (BMS-963272) Dosing Regimen 1 (Experimental)
  Interventions: Drug: BMS-963272
- Active Treatment (BMS-963272) Dosing Regimen 2 (Experimental)
  Interventions: Drug: BMS-963272
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo matching BMS-963272

INTERVENTIONS:
Drug: BMS-963272 — Specified dose on specified days
  Arms: Active Treatment (BMS-963272) Dosing Regimen 1; Active Treatment (BMS-963272) Dosing Regimen 2
Other: Placebo matching BMS-963272 — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and drug levels of BMS-963272 compared to placebo in participants with nonalcoholic fatty liver disease (NAFLD) and high probability of advanced fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 30 kg/m^2
* Magnetic resonance imaging-proton density fat fraction (MRI-PDFF) ≥ 10% as evaluated by central review
* FibroScan-based transient elastography ≥ 9.9 kPa
* Alanine aminotransferase (ALT): > 30 U/L
* If available, historical diagnosis of non-alcoholic steatohepatitis (NASH) according to NASH Clinical Research Network classification by liver biopsy within 6 months before screening will be recorded
* Must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Women who are breastfeeding
* Inability to tolerate the mixed meal or the testing conditions, oral medication, venipuncture and/or inadequate venous access
* History or current diagnosis of cirrhosis, hepatocellular carcinoma (HCC), or hepatic decompensation
* Recent history (within 2 years before screening) of drug or alcohol abuse or excessive alcohol intake, defined as 30 g/day (men) or 20 g/day (women)
* Use of lipase inhibitors such as orlistat within 4 weeks before screening or during screening
* Use of glucagon-like peptide-1 (GLP-1) receptor agonists within 12 weeks before screening or during screening
* Uncontrolled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg) during screening, unless discussed with the Medical Monitor
* Glycated hemoglobin (HbA1c) ≥ 9.5%
* NASH-modifying therapies including investigational therapies (e.g., obeticholic acid, ursodeoxycholic acid) within 90 days before screening or during screening
* Medications for obesity within 12 weeks before screening, or during screening
* If taking vitamin E at a dose ≥ 800 mg/day, the dose must be stable beginning at least 6 months before screening and should remain stable during screening
* If taking a thiazolidinedione, the dose must be stable beginning at least 12 weeks before screening and should remain stable during screening
* If taking a dipeptidyl peptidase (DPP)-4 inhibitor or other medications for diabetes, the dose must be stable beginning at least 12 weeks before screening and should remain stable during screening
* If taking insulin, the dose may be altered by up to 10% within 12 weeks before screening and during the screening period
* If taking a statin or other prescription or over-the-counter lipid-lowering drug, the dose must be stable beginning at least 6 weeks before screening and should remain stable during screening

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 166 days
Incidence of serious adverse events (SAEs) | Up to 166 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 166 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 166 days
Incidence of clinically significant changes in physical examination findings | Up to 166 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 166 days
  PR interval: The time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS interval | Up to 166 days
  QRS interval: A combination of the Q wave, R wave and S wave, the "QRS complex" represents ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 166 days
  QT interval: Measured from the beginning of the QRS complex to the end of the T wave
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF interval | Up to 166 days
  QTcF interval: Corrected QT interval using Fridericia's formula (QTcF)
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry test | Up to 166 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 166 days
Incidence of clinically significant changes in clinical laboratory results: Coagulation tests | Up to 166 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 46 days
Incidence of clinically significant changes in clinical laboratory results: Liver function tests | Up to 166 days
Incidence of clinically significant changes in clinical laboratory results: Lipid panel tests | Up to 166 days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) sampling: Maximum observed plasma concentration (Cmax) | Day 1 and Day 84
Pharmacokinetic (PK) sampling: Time to maximum observed plasma concentration (Tmax) | Day 1 and Day 84
Pharmacokinetic (PK) sampling: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Day 1 and Day 84
Trough observed plasma concentration (Ctrough) | Day 1, Day 15, Day 29, Day 57, and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (18):
  - Cullman Clinical Trials, Cullman, Alabama
  - Local Institution, Chandler, Arizona
  - Arizona Liver Health - Tucson, Tucson, Arizona
  - Local Institution, Boca Raton, Florida
  - RecioMed Clinical Research Network, Boynton Beach, Florida
  - Local Institution, Miami, Florida
  - Advanced Pharma - Miami, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Local Institution, Port Orange, Florida
  - Local Institution, Bastrop, Louisiana
  - Local Institution, Biloxi, Mississippi
  - Local Institution, Kansas City, Missouri
  - Local Institution, Chattanooga, Tennessee
  - Local Institution, Germantown, Tennessee
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - Local Institution, Edinburg, Texas
  - Local Institution, McAllen, Texas
  - Local Institution, San Antonio, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm